CLINICAL TRIAL: NCT05494944
Title: Low Power Thulium Enucleation of Prostate More Than 80 Grams
Brief Title: Low Power ThULEP for Prostate Size More Than 80 gm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Lecturer, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Urology department
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ThuLEP group (Other)
  Interventions: Procedure: ThuLEP

INTERVENTIONS:
Procedure: ThuLEP — Minimal invasive prostate intervention

SUMMARY:
Feasibility and Efficacy of lower power thulium enucleation of prostate more than 80 grams

DETAILED DESCRIPTION:
Intra operative outcome and postoperative follow up of IPSS score and IEFF score at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BPH patients with failed medical treatment
* Refractory retention
* Hematuria
* Bladder stones
* Renal impairment due to BPH

Exclusion Criteria:

* Neurogenic patients
* stricture urethra

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Timing of complete adenoma removal ( enucleation time in minutes) | During operation
International prostate symptoms score IPSS less than 7 which is good outcome | 12 months

SECONDARY OUTCOMES:
International Index of Erectile Function- 5 score more than 12 which is a good outcome | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samer Morsy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morsy S, Kamal I, Meshref A, Abdel-Mohsen M, Abdel-Hakim M, Yehia A. Surgical outcomes of low-power thulium laser enucleation of prostates >80 g. One-year of follow-up. Cent European J Urol. 2023;76(3):193-198. doi: 10.5173/ceju.2023.50. Epub 2023 Jul 12. PMID 38045774